CLINICAL TRIAL: NCT00005934
Title: A Pilot Study of 5-Azacytidine and Oral Sodium Phenylbutyrate in Severe Thalassemia
Brief Title: 5-Azacytidine and Phenylbutyrate to Treat Severe Thalassemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000166; 00-DK-0166; NCT00007072 (obsolete NCT alias)
Record Dates: First submitted 2000-07-06; First posted 2000-07-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-06

CONDITIONS: Beta Thalassemia
Keywords: Fetal Hemoglobin; 5-Azacytidine; Phenylbutyrate; Thalassemia; Hemoglobin; Anemia; Blood; Thalassemia Major; Beta Thalassemia
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Anemia | interventions — Azacitidine

INTERVENTIONS:
Drug: 5-Azacytidine

SUMMARY:
This study will evaluate the safety and effectiveness of 5-azacytidine and phenylbutyrate for treating thalassemia major. Patients with this disease have abnormal production of hemoglobin (the oxygen-carrying protein in red blood cells), which leads to red blood cell destruction. As a result, patients require frequent red cell transfusions over many years. Because of these transfusions, however, excess iron is deposited in various body organs-such as the heart, liver, thyroid gland and, in men, the testes-impairing their function.

Fetal hemoglobin-a type of hemoglobin that is produced during fetal and infant life-can substitute for adult hemoglobin and increase the levels of red cells in the body. After infancy, however, this type of hemoglobin is no longer produced in large quantities. 5-azacytidine can increase fetal hemoglobin levels, but this drug can damage DNA, which in turn can increase the risk of cancer. This study will try to lessen the harmful effects of 5-azacytidine by using only one or two doses of it, followed by long-term therapy with phenylbutyrate, a drug that may be as effective as 5-azacytidine with less harmful side effects.

Patients 18 years of age and older with severe thalassemia major may be eligible for this study. Before beginning treatment, candidates will have a medical history and physical examination, blood tests, chest X-ray, electrocardiogram (EKG), bone marrow biopsy (removal of a small sample of bone marrow from the hip for microscopic examination) and whole-body magnetic resonance imaging (MRI). For the biopsy, the area of the hip is anesthetized and a special needle is inserted to draw bone marrow from the hipbone. For the MRI scan, a strong magnetic field is used to produce images that will identify sites where the body is making red blood cells. During this procedure, the patient lies on a table in a narrow cylinder containing a magnetic field. Earplugs are placed in the ears to muffle the loud thumping sounds the machine makes when the magnetic fields are being switched.

An intravenous (IV) catheter (flexible tube inserted into a vein) is placed in a large vein of the patient's neck, chest or arm for infusion of 5-azacytidine at a constant rate over 4 days. Patients who do not respond to this first dose of 5-azacytidine will be given the drug again after about 50 days. If they do not respond to the second dose, alternate treatments will have to be considered. Patients who respond to 5-azacytidine will begin taking phenylbutyrate on the 14th day after 5-azacytidine was started. They will take about 10 large pills 3 times a day, continuing for as long as the treatment is beneficial. All patients will be hospitalized for at least 6 days starting with the beginning of 5-azacytidine therapy. Those who are well enough may then be discharged and continue treatment as an outpatient.

Patients will be monitored with blood tests daily for 2 weeks and then will be seen weekly for about another 5 weeks. Bone marrow biopsies will be repeated 6 days after treatment begins and again at 2 weeks and 7 weeks. MRI will be repeated 7 weeks after treatment begins. After 7 weeks, patients will be seen at 3-month intervals. Bone marrow biopsies will be done every 6 months for the first 3 years after treatment. Patients will have red cell transfusions as needed and chelation therapy to remove excess iron.

DETAILED DESCRIPTION:
Individuals with homozygous beta-thalassemia are either severely anemic or dependent on blood transfusion to sustain life. Deficient synthesis of the beta chain leads to imbalanced chain synthesis with an excess of alpha globin. This alpha globin precipitates, causing ineffective erythropoiesis and shortened red cell survival. In patients with homozygous beta-thalassemia, enhanced gamma globin synthesis could partially compensate for the deficient synthesis of beta globin rendering chain synthesis more balanced and reducing the relative excess of alpha chains. The purpose of this protocol is to test the hypothesis that induction therapy with 5-azacytidine, followed by maintenance treatment with oral phenylbutyrate will enhance gamma globin synthesis, increase red cell production and partially or substantially correct the anemia in patients with homozygous beta-thalassemia.

ELIGIBILITY:
INCLUSION CRITERIA:

Thalassemia major with progressive disease or complications of iron overload despite traditional transfusion and iron chelation therapy

Thalassemia major in which standard transfusion therapy or iron chelation therapy is contraindicated

ECOG performance status must be less than or equal to 2

NYHA less than or equal to class II status

Progressive disease is defined as 1) an increasing transfusion requirement or difficulty in maintenance of hemoglobin levels greater than 7g/dl as a consequence of autologous or allogeneic antibodies or 2) increasing extramedullary hematopoiesis causing compression phenomena.

Complications of iron overload despite iron chelation therapy is defined as difficulty in achieving negative iron balance when complications of iron overload exist. Complications of iron overload include heart failure, or decreased cardiac ejection fraction, endocrinopathy and evidence of progressive liver dysfunction.

EXCLUSION CRITERIA:

Severe sepsis or septic shock

Current pregnancy or breast feeding

Not able to give informed consent

Altered mental status or seizure disorder

AST or ALT greater than 3X upper limit of normal

Bilirubin greater than1.5X upper limit of normal, unless the abnormal bilirubin can be accounted for by indirect hyperbilirubinemia due to hemolysis or Gilbert's Disease

Serum albumin less than 3g/dl

Creatinine greater than 2mg/dl and creatinine clearance less than 60ml/min

Patients who are moribund or patients with concurrent hepatic, renal, cardiac, metabolic, or any disease of such severity that death within 7-10 days is likely

Concurrent myelodysplastic syndrome or leukemia

NYHA class III/IV status

ECOG performance status greater than 2

Age less than 18 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Start 2000-06; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Thomas ED, Buckner CD, Sanders JE, Papayannopoulou T, Borgna-Pignatti C, De Stefano P, Sullivan KM, Clift RA, Storb R. Marrow transplantation for thalassaemia. Lancet. 1982 Jul 31;2(8292):227-9. doi: 10.1016/s0140-6736(82)90319-1. No abstract available. PMID 6124668
- [Background] Wolfe L, Olivieri N, Sallan D, Colan S, Rose V, Propper R, Freedman MH, Nathan DG. Prevention of cardiac disease by subcutaneous deferoxamine in patients with thalassemia major. N Engl J Med. 1985 Jun 20;312(25):1600-3. doi: 10.1056/NEJM198506203122503. PMID 4000198
- [Background] Modell B, Petrou M. Management of thalassaemia major. Arch Dis Child. 1983 Dec;58(12):1026-30. doi: 10.1136/adc.58.12.1026. No abstract available. PMID 6660889